CLINICAL TRIAL: NCT06538168
Title: The Effect of a Comprehensive Digital Health Education on Self-Foot Care and Quality of Life Among Patients With Diabetes
Brief Title: Effectiveness of a Digital Health Education on Self-Foot Care and Quality of Life Among Patients With Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Collaborators: University of Lahore (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD studentship, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: UIPH
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: In an interventional parallel study design, participants are assigned to either an intervention group and a control group. The intervention group receives the treatment or intervention being tested, while the control group does not receive the intervention and serves as a comparison. This allows researchers to assess the effectiveness of the intervention by comparing outcomes between the two groups under controlled conditions.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and/or assessors are unaware of who receives the intervention (treatment) or control. This reduces bias by ensuring that knowledge of the treatment does not influence outcomes assessment, thus enhancing the reliability of study results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group typically consists of participants who are subjected to the Diabetes Self-Management Education (DSME) program The intervention, Diabetes Self-Management Education (DSME), involves a structured educational program including daily reminders regarding medication, and foot care, educational-led video weekly, and handouts for the management of diabetes and foot care to enhance knowledge and skills in managing diabetes and preventing complications like diabetic foot ulcers (DFUs).
  Interventions: Behavioral: Diabetes Self-Management Education (DSME)
- Control group (No Intervention): These participants do not receive any intervention.

INTERVENTIONS:
Behavioral: Diabetes Self-Management Education (DSME) — The intervention, Diabetes Self-Management Education (DSME), involves a structured educational program including daily reminders regarding medication, and foot care, educational-led video weekly, and handouts for the management od diabetes and foot care to enhance knowledge and skills in managing diabetes and preventing complications like diabetic foot ulcers (DFUs).
  Arms: intervention group

SUMMARY:
Diabetes is a significant global health concern, affecting over half a billion people and leading to severe complications like diabetic foot ulcers (DFUs). The increasing incidence of DFUs highlights the need for ongoing research and effective prevention strategies. A major challenge in managing DFUs is the inadequate preparation of healthcare professionals (HCPs) in delivering comprehensive diabetes self-management education (DSME). Enhancing the education and training of HCPs is essential to improve diabetes management and reduce DFUs.

Studies show that patients' knowledge and self-care practices vary widely, with common foot-care activities including washing, drying, applying moisturizer, and routine nail care. Improving these self-care practices is crucial for early recognition and management of DFUs to reduce the risk of amputations.

Health promotion models such as the Self-Efficacy Theory and Health Belief Model have shown promise in informing foot care interventions, but further research is needed to determine the most effective strategies. Previous research has several limitations, including selection bias, lack of consensus on outcome measures, and moderate risk of bias in some studies.

The proposed study will use an experimental design with a nonequivalent control group to assess the effectiveness of DSME in reducing non-ulcerated diabetic foot incidents. Data will be collected using the Diabetes Self-Care Activities Foot Care Questionnaire and analyzed with statistical tests. Ethical guidelines will be strictly followed, ensuring participant confidentiality and voluntary participation.

Overall, this research aims to address gaps in diabetes education and promote behavioral changes to improve diabetes care and reduce DFUs. Continuous training and education for HCPs are vital for enhancing their competence in managing DFUs and improving patient outcomes.

DETAILED DESCRIPTION:
Diabetes is a major global health issue affecting over half a billion people worldwide, leading to serious complications such as diabetic foot ulcers (DFUs). The increasing incidence of DFUs necessitates further research to manage and prevent these severe complications. Healthcare professionals (HCPs) play a crucial role in addressing the rising incidence of diabetes and DFUs through capacity building and periodic education. However, many HCPs are inadequately prepared to deliver comprehensive diabetes self-management education (DSME), which is essential for preventing and treating DFUs.

The World Health Organization (WHO) reports that approximately 422 million people with diabetes live in low- and middle-income countries, with diabetes directly causing about 1.5 million deaths annually. Over the past few decades, there has been a consistent rise in both the incidence and prevalence of diabetes. This condition significantly contributes to renal disease, heart attacks, strokes, blindness, and lower extremities amputation, often resulting from infected foot ulcers. About 15% to 25% of diabetic patients develop foot ulcers at some point. Foot problems like ulcers, infections, and amputations are among the most significant complications of diabetes, but these issues can often be avoided with consistent foot care.

The study aims to understand how health promotion models have informed foot care interventions for older adults with diabetes. A review of 2,078 articles identified 31 studies that met eligibility criteria, focusing on foot care interventions for older adults. Most of these studies involved people with diabetes and used health promotion models such as the Self-Efficacy Theory and the Health Belief Model. The interventions showed promising outcomes in improving foot care for older adults, highlighting the need for further research to determine the most effective models and implementation strategies.

Previous research has several limitations: exclusion of relevant studies on intervention implementation, lack of consensus on foot-related outcome measures, selection bias due to convenience sampling techniques, cross-sectional designs making causal inferences impossible, moderate risk of bias in some studies, restriction to studies conducted between 2004 and 2022, lack of randomized or controlled samples in some studies, and immediate assessment of attitudes and skills post-training influencing health promotion models.

This research addresses the lack of diabetes education and the limited adoption of behavioral changes among the population, which lead to challenges in diabetes care. Effective education for healthcare professionals, communities, and patients is essential to improve diabetes management and reduce the risk of complications such as DFUs. The objectives of the study are to understand the contexts where health promotion models have informed foot care interventions, identify the health promotion models used in these interventions, and document the effectiveness of theoretically informed health promotion interventions in improving foot care for older adults.

Health promotion models like the Self-Efficacy Theory and the Health Belief Model have shown promising outcomes in improving foot care behaviors and knowledge. The studies vary in intervention approaches, delivery methods, and outcome measurements, emphasizing the need for further research to determine the most effective models and implementation strategies. There is a strong correlation between high knowledge of foot care and good practice, with varying levels of knowledge and engagement in foot-care activities like washing, drying, applying moisturizer, and trimming nails.

The study will assess the impact of DSME on non-ulcer diabetic foot incidents through a structured research design and statistical analysis. A review of existing studies shows that appropriate foot care practices are essential for preventing complications like DFUs. Common self-care practices include washing feet with lukewarm water, drying thoroughly, using moisturizing cream, inspecting feet daily, nail care, and wearing suitable footwear. Outcome measures in these studies included foot health outcomes, knowledge of foot health, foot care behaviors, and self-efficacy. The need for standardized outcome measures and further research on the effectiveness and cost-benefit of foot care interventions for older adults is highlighted.

The study will use an experimental design with a nonequivalent control group. Consecutive sampling will divide 230 participants into intervention and control groups. The Diabetes Self-Care Activities Foot Care Questionnaire will be used as the research instrument. Statistical analyses will include the Wilcoxon Signed Ranks Test and Mann-Whitney Test to compare the mean incidence of non-ulcerated diabetic foot incidents before and after the intervention.

The research will adhere to ethical guidelines, ensuring participant confidentiality, voluntary participation, and informed consent. Participants will be assured of their right to withdraw from the study at any time without any penalties.

Overall, this research aims to enhance diabetes education and promote behavioral changes to improve diabetes care and reduce the incidence of DFUs. Continuous training and education for HCPs are crucial for improving their competence in managing DFUs and achieving better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a diabetic foot wound corresponding to Warner 2 - 4 Continuous existence of the diabetic foot lesion for a minimum of 4 weeks < Participant has given written informed consent

Exclusion Criteria:

* Age <18 years Pregnancy Present or expected non-compliance with the requirements of the study estimated by investigator at the time point of inclusion indication for amputation above the ankle level of the same Necrotic tissue with eschar present that cannot be debrided untreated osteitis or osteomyelitis Unexplored fistula

  * Malignancy of the wound Exposed nerves, vessels, or anastomotic areas
  * Ambulant negative pressure wound therapy of patients with anticoagulation therapy or higher grade impaired clotting function and a heightened risk for bleeding with relevant circulatory effects
  * Allergy to any disposal component of each treatment arm Severe anemia which is not caused by an infection
  * Simultaneous participation in other interventional trials / previous participation in this trial
  * Use of negative pressure wound therapy within 6 weeks before randomization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2430 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Diabetic foot | 12 months from baseline
  Knowledge of Diabetic foot using a scale will be measured Likert Scale questions where participants rate their agreement with statements about foot care practices (e.g., "I always wear well-fitting shoes," with options ranging from "Strongly Disagree" to "Strongly Agree").
  The total score is then used to categorize the participant's knowledge level. This categorization can be study-specific, but some common examples include:
  * Low knowledge: Scoring less than 60% of questions correctly suggests a need for significant education on diabetic foot care.
  * Moderate knowledge: Scoring between 60% and 80% indicates some understanding but may benefit from further education.
  * High knowledge: Scoring above 80% suggests a good understanding of diabetic foot care principles.
Health related quality of life | 12 months from baseline
  Health related quality of life measured by EQ- 5D-3L. o measure the health-related quality of life at baseline, three-month, and 12-month post-intervention, EuroQol 5-Dimension- 3-level will be used. The European quality of life scale (EQ-5D-3L) has five dimensions and three levels. Each of the five dimensions comprising the EQ-5D descriptive system is divided into three levels of perceived problems: LEVEL 1: indicating no problem LEVEL 2: indicating some problems LEVEL 3: indicating extreme problems, 1 (perfect health), with higher scores indicating higher health utility.
  2- On a 20 cm vertical visual analog scale, the EQ-VAS captures the patient's self-rated health, with two unique endpoints such as "Best imaginable health condition" for a score of 100 and "Worst imaginable health state" for a score of 0.
Adherence to anti-diabetic medication | 12 months from baseline
  The secondary outcome is the change in medication adherence to antihypertensive treatment. Using the "pills taken over a certain period, divided by pills prescribed for that specific period", the primary outcome will be measured.it will be self-reporting. A cut-off value of 80% has been established from previous literature. Non-adherents will make up less than 80% of the population, while adherents will make up more than 80%.

SECONDARY OUTCOMES:
Past 3 months glycemic control | 12 months from baseline
  The out come will be measured by HbA1c
Hospitalization | 12 months from baseline
  measured by tracking for hospital admission
Amputation status | 12 months from baseline
  Amputation status measured by confirming hospital records
Foot ulceration | 12 months from baseline
  Foot ulceration will be measured by Wagner Wound Classification System Wagner Grade 0: Skin is intact with no open lesion or a pre-ulcerative lesion - may have a deformity or cellulitis Wagner Grade 1: Partial- or full-thickness ulcer (superficial ulcer) Wagner Grade 2: Deep ulcer extended to ligament, tendon, joint capsule, bone, or deep fascia without abscess or osteomyelitis (OM) Wagner Grade 3: Deep abscess, OM, or joint sepsis Wagner Grade 4: Partial-foot gangrene Wagner Grade 5: Whole-foot gangrene

REFERENCES:
- [Result] Ackermann RT, O'Brien MJ. Evidence and Challenges for Translation and Population Impact of the Diabetes Prevention Program. Curr Diab Rep. 2020 Feb 20;20(3):9. doi: 10.1007/s11892-020-1293-4. PMID 32080770
- [Result] Arumalla N, Chan CKD, Gibson M, Man YL, Adas MA, Norton S, Galloway JB, Garrood T. The Clinical Impact of Electronic Patient-Reported Outcome Measures in the Remote Monitoring of Inflammatory Arthritis: A Systematic Review and Meta-analysis. Arthritis Rheumatol. 2023 Nov;75(11):1892-1903. doi: 10.1002/art.42559. Epub 2023 Sep 18. PMID 37204273
- [Result] Geidne S, Kokko S, Lane A, Ooms L, Vuillemin A, Seghers J, Koski P, Kudlacek M, Johnson S, Van Hoye A. Health Promotion Interventions in Sports Clubs: Can We Talk About a Setting-Based Approach? A Systematic Mapping Review. Health Educ Behav. 2019 Aug;46(4):592-601. doi: 10.1177/1090198119831749. Epub 2019 Feb 22. PMID 30795690
- Available data/document: Informed Consent Form — https://www.facebook.com/gghgmabadfsd/?paipv=0&eav=AfbwgEmoehvAkH8F8E-KZ9WClHEgcLyNQwBOij0PYLNHpvrJZ1KZbTJdZYuWB21J8rA&_rdr